CLINICAL TRIAL: NCT05201183
Title: A Dose Escalation Study of Intensity Modulated Total Marrow Irradiation (IMRT-TMI) Followed by Fludarabine as a Myeloablative Conditioning Regimen for Allogeneic Hematopoietic Stem Cell Transplantation for Patients With Relapsed and Refractory Hematologic Malignancies
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: insufficient staff and updates in standard practice have made it difficult to recruit participants
Sponsor: Naoyuki G. Saito, M.D., Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Naoyuki G. Saito, M.D., Ph.D., Assistant Professor of Radiation Oncology, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTO-IUSCCC-0747
Record Dates: First submitted 2022-01-07; First posted 2022-01-21 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Acute Myeloid Leukemia; Chronic Myeloid Leukemia; Acute Lymphocytic Leukemia; Myelodysplastic Syndromes
Keywords: Radiation; Total Marrow Irradiation; Fludarabine; Bone Marrow Transplant
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes | interventions — fludarabine

STUDY DESIGN:
Intervention Model Description: A standard "3+3" phase I design of dose escalation using 3 patients per dose level cohort with an expansion to 6 patients at the MTD will be used in Phase I. We will treat 3 patients at the initial dose level of TMI. If no dose-limiting toxicity (DLT) is observed, the next cohort of three patients is treated at the next higher dose level. If 1 of the 3 patients demonstrates DLT, an additional 3 patients are treated at that dose level. If only 1 of the 6 shows DLT, the next cohort of three patients is entered at the next dose level. If 2 or more of the 6 demonstrate DLT, the MTD is defined as the previous dose level. If no DLT is observed in the final dose level, the number of patients treated will be expanded to 6. In phase II, we will enroll additional patients at the defined MTD level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Fludarabine + Total Marrow Irradiation (Experimental): Fludarabine will be administered sequentially after the administration of TMI. TMI will be delivered on Days -11, -10, -9, -8, and -7 (1.4-2.2 gray (GY)/fraction, twice a day) followed by fludarabine on Days -6, -5, -4, -3, and -2 (150 mg/m2, 30 mg/m2/day)
  Interventions: Combination Product: Fludarabine + Total Marrow Irradiation

INTERVENTIONS:
Combination Product: Fludarabine + Total Marrow Irradiation — Patients will receive total marrow irradiation TMI on Day -11 to Day -7 in two fractions per day. The TMI dose will be escalated in successive cohorts compromised of 3-6 patients as follows:
  Cohort 1 1.4 (Gy/fraction) Cohort 2: 1.6 (Gy/fraction) Cohort 3 1.8 (Gy/fraction) Cohort 4 2.0 (Gy/fraction) Cohort 5 2.2 (Gy/fraction)
  Patients will receive Fludarabine (30 mg/m2/day) on Day -6 to Day -2 followed by allo-HSCT on Day 0.

SUMMARY:
This is a phase I/II clinical trial to determine the maximum tolerated dose (MTD) of total marrow irradiation (TMI) followed by fludarabine in the context of a myeloablative conditioning regimen for allogeneic hematopoietic stem cell transplantation (allo-HSCT), as well as to determine the efficacy of the regimen in patients with high-risk leukemia and myelodysplasia.

DETAILED DESCRIPTION:
This is a phase I/II clinical trial to determine the maximum tolerated dose (MTD) of total marrow irradiation (TMI) followed by fludarabine in the context of a myeloablative conditioning regimen for allogeneic hematopoietic stem cell transplantation (allo-HSCT), as well as to determine the efficacy of the regimen in patients with high-risk leukemia and myelodysplasia. TMI, which allows for conformal dosing of target bone marrow tissue while giving lower doses to organs at risk, is considered by many to be a superior alternative to conventional total body irradiation (TBI). Through the use of TMI, it is possible to escalate the dose of radiation to the bone marrow while keeping the dose to normal organs at acceptable levels, effectively widening the therapeutic window of this modality. This conditioning regimen will be tried in patients with relapsed or refractory hematologic malignancies.

Primary Objectives:

Phase I: Determine the MTD of TMI (delivered twice a day for 5 days) followed by fludarabine (fixed at 150 mg/m2 given over 5 days) as a conditioning regimen for Allo-HSCT for patients with high risk (relapsed/refractory) acute lymphocytic leukemia (ALL), acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), and chronic myelogenous leukemia (CML).

Phase II: Single-arm exploratory study to expand the cohort at the MTD level to estimate 1- year overall survival (OS), with the objective of increasing the OS from the historical rate of 30% (null hypothesis) to 50% (alternate hypothesis) with 80% power and a one-sided type I error of 0.05.

Secondary Objectives

1. Describe the extramedullary toxicity and the incidence of complications, including mucositis, acute and chronic graft versus host disease (GvHD), sinusoidal obstruction syndrome (SOS), and pneumonitis.
2. Describe the time to engraftment of neutrophils and platelets
3. Describe the disease response rate at Day 30 after transplantation
4. Describe the overall survival and disease-free survival
5. Describe the cumulative incidence of relapse and non-relapse mortality 6
6. Determine the correlation between plasma/serum markers and radiation induced acute and long term toxicities.
7. Describe the quality of life metrics of participating subjects

ELIGIBILITY:
Inclusion Criteria:

1. Documentation of Disease: Patients must be diagnosed with one of the following conditions:

   1. Acute Myeloid Leukemia (AML), with no history of extramedullary disease, who are not in complete remission, who have either primary refractory or relapsed disease, and who do not have more than one of the following adverse factors:

      * Duration of first CR < 6 months (if previously in CR), based on the best overall clinical assessment of the disease course, not solely based on blood test or bone marrow biopsy results
      * Poor risk karyotype including any of the following: complex karyotype with ≥3 clonal abnormalities, 5q-/-5, 7q-/-7, 11q23 abnormalities, inv(3q), 20q or 21q abnormalities, t (6;9), t (9;22), 17p abnormalities [or TP53 mutations] or monosomal karyotype. Molecular typing (except for TP53 mutation) will not be used for eligibility criteria determination.
      * Circulating peripheral blood blasts at time of enrollment
      * Karnofsky performance status <90%
   2. Acute Lymphocytic Leukemia (ALL) who are not in complete remission, who have either primary refractory or relapsed disease, and who do not have more than one of the following adverse factors:

      * Primary refractory or first relapse. Patients in second or subsequent relapse are excluded.
      * Bone marrow blasts >25% within 30 days before the start of the conditioning regimen
      * Age >40 years
   3. Myelodysplasia with a Revised International Prognostic Score (IPSS-R) of greater than 4.5 (i.e., high- or very-high risk).
   4. Chronic Myelogenous Leukemia (CML) in accelerated phase, defined by any of the following:

      * 10-19% blasts in peripheral blood white cells or bone marrow
      * Peripheral blood basophils at least 20%
      * Persistent thrombocytopenia (< 100 x 109/l) unrelated to therapy, or persistent thrombocytosis (>1000 x 109/l) unresponsive to therapy
      * Increasing spleen size and increasing white blood cell (WBC) count unresponsive to therapy
      * Cytogenetic evidence of clonal evolution (i.e., the appearance of an additional genetic abnormality that was not present in the initial specimen at the time of diagnosis of chronic phase)
2. The patient must be 18-65 years old at time of consent
3. Signed written informed consent: Patient must be capable of understanding the investigational nature of this study, potential risks and benefits of the study, and be able to provide a valid informed consent.
4. Availability of a consenting human leukocyte antigens (HLA)-matched donor
5. Karnofsky Performance Status 70% or higher
6. Required baseline laboratory values:

   * Estimated creatinine clearance ≥ 60 ml/min
   * Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x upper limit of normal value
   * Bilirubin ≤ 1.5 x upper limit of normal value (unless determined to be related to Gilbert's disease)
7. Required baseline cardiac function values:

   * Required baseline cardiac function of left ventricular ejection fraction (LVEF) > 45 % corrected
8. Required baseline pulmonary function values:

   * Required baseline pulmonary function of lung diffusing capacity (DLCO) > 45 % predicted (corrected for hemoglobin))

Exclusion Criteria:

1. HIV seropositive patients
2. Pregnant or nursing females.
3. Prior radiation therapy
4. Patients who have had a prior autologous or allogeneic bone marrow or stem cell transplantation
5. Gemtuzumab ozogamicin (trade name: Mylotarg) and/or inotuzumab ozogamicin (trade name: Besponsa) use within 60 days before start of the conditioning regimen
6. Though this is NOT an exclusion criterion, we strongly recommend discontinuation of any steroidal oral contraceptives at least 7 days before start of the conditioning regimen. Use of therapeutic alternatives, including leuprolide should be considered to reduce the risk of SOS/VOD. Of note, for patients already on steroidal oral contraceptives for excessive menorrhagia, the switch to leuprolide should occur at least 2 weeks before the start of the conditioning regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of Total Marrow Irradiation (TMI) followed by 150 mg/m2 fludarabine- Phase I only | Day -10 of conditioning regimen through 30 days post transplant (40 days)
Overall survival (OS) rate 1 year post transplant-Phase II only | 1 year

SECONDARY OUTCOMES:
Frequency of non hematologic toxicity | 100 days
Incidence of mucositis | 100 days
Incidence of acute graft versus host disease | 100 days
Incidence of chronic graft versus host disease | 100 days
Incidence of sinusoidal obstruction syndrome | 100 days
Incidence of pneumonitis | 100 days
Time to engraftment of neutrophils | rom date of transplant to the first of three consecutive days after transplantation during which the absolute neutrophil count (ANC) is greater than or equal to 0.5 x 10^9/liter
Time to engraftment of platelets | the time from Day 0 to the first of seven consecutive days after transplantation during which the platelet count is at least 20 x109/l without transfusion support.
Disease free survival | 3 years
Mean Quality of Life (QOL) as measured by Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) version 4 | At screening, Day +30, Day +180, Day +365, Day +730 and Day +1095 from transplant (approximately 3 years)
  50 item likert type scale with responses measuring from 0-4 (where 0 = not at all; 1 = a little bit; 2 = somewhat, 3 = quite; and 4 = very much) with higher scores correlating to higher QOL
Incidence of non-relapse mortality | 30 days
Incidence of non-relapse mortality | 100 days
Incidence of non-relapse mortality | 1 year
Incidence of relapse mortality | 1 year
Incidence of relapse mortality | 30 days
Incidence of relapse mortality | 100 days
Overall Survival | Day +30, Day +100 and 1 year (approximately 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Naoyuki Saito, MD PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No